CLINICAL TRIAL: NCT04455971
Title: A Naturalistic, Longitudinal, Observational Study of Associations Between Frequency of Orgasmic Meditation Practice, Occurrence of Female Physiological Orgasm and Sleep Quality
Brief Title: Orgasmic Meditation and Sleep Quality
Status: Completed | Type: Observational
Sponsor: Institute of OM Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: OMSLEEP
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Sleep

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OM Group: People who participate in the practice of orgasmic meditation (OM)
  Interventions: Behavioral: Orgasmic Meditation

INTERVENTIONS:
Behavioral: Orgasmic Meditation — Orgasmic Meditation (OM) is a form of meditation that increases bodily awareness during structured, partnered female genital stimulation over a 15-minute period.

SUMMARY:
The primary purpose of this study is to use an observational design to examine whether the practice of orgasmic meditation (OM) is associated with app-based measures of sleep quality. A secondary purpose of this study is to examine whether the occurrence of physiological orgasm during OM practice is associated with app-based measures of sleep quality. It is hypothesized that the practice of OM will have a positive impact on sleep quality.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, males and females, no exclusion by race, ethnicity or sexual orientation
2. Experienced in OM practice ("experienced" defined as >10 OM sessions in lifetime)
3. Currently practicing OM and participating in ≥1 OM session per week on average
4. Willingness to calibrate the Sleep Cycle app and use it for 30 continuous nights
5. Ability to charge phone by bed overnight during sleep
6. Ability to place phone near the bed, such as on a nightstand table overnight during sleep

Exclusion Criteria:

1. Inability to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Correlation between sleep quality and occurrence and frequency of OM sessions during the prior day | 30 days
  "Sleep quality" will be measured using the Sleep Cycle app

SECONDARY OUTCOMES:
Correlation between sleep duration and occurrence and frequency of OM sessions during the prior day | 30 days
  "Sleep duration" will be measured using the Sleep Cycle app
Correlation between time to fall asleep and occurrence and frequency of OM sessions during the prior day | 30 days
  "Time to fall sleep" will be measured using the Sleep Cycle app
Correlation between sleep regularity and occurrence and frequency of OM sessions during the prior day | 30 days
  "Sleep regularity" will be measured using the Sleep Cycle app
Change in total sleep duration during nights following OM and nights following no OM | 30 days
  "Sleep duration" will be measured using the Sleep Cycle app
Change in time to fall asleep during nights following OM and nights following no OM | 30 days
  "Time to fall sleep" will be measured using the Sleep Cycle app
Change in sleep regularity during nights following OM and nights following no OM | 30 days
  "Sleep regularity" will be measured using the Sleep Cycle app

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raison, MD, Principal Investigator — Institute of OM Foundation
Locations (1):
- Institute of OM Foundation, Santa Rosa, California, United States

IPD SHARING:
Plan to Share IPD: No